CLINICAL TRIAL: NCT00486057
Title: A Retrospective Review of Daclizumab Experience in Pediatric Heart Transplant
Brief Title: Daclizumab Experience in Pediatric Heart Transplant
Status: Terminated | Type: Observational
Why Stopped: sufficient data collected for conclusion of retrospective study
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Director Research, Children's Healthcare of Atlanta Institutional Review Board
Other Study IDs: 06-199
Record Dates: First submitted 2007-06-12; First posted 2007-06-13 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2007-11

CONDITIONS: Congenital Disorders
Keywords: Daclizumab; Immuno-suppression protocol; Heart Transplant; Rejection
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Rejection, Psychology

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to examine the outcomes of those who have received Daclizumab as part of their immuno-suppression protocol following heart transplantation. Literature suggests that the time to first rejection episode can be avoided or delayed by using induction therapy.

DETAILED DESCRIPTION:
In August 2005 the heart transplant team at Children's Healthcare of Atlanta began a protocol of Daclizumab 1mg/kg IV every two weeks for 5 doses; 1st dose to be received in the operating room following discontinuation of cardiopulmonary bypass.

Since one year has passed following initiation of this practice, it is necessary to review this immuno-suppression strategy and determine if, in fact, there was clinical benefit of reducing rejection without increasing the vulnerabilities of the immuno-compromised host.

We wish to review all heart transplant recipient records between August 1, 2004 and October 15, 2006. Historically, Children's has done approximately 10 transplants per year; therefore, we will review approximately 15 charts at Children's Healthcare of Atlanta and Sibley Heart Center Cardiology.

ELIGIBILITY:
Inclusion Criteria:

* Status post heart transplant
* Age 0-21 years
* Received Daclizumab as induction therapy

Exclusion Criteria:

* Those who do not meet inclusion criteria

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Status post heart transplant Age 0-21 years Received Daclizumab as induction therapy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2004-08; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirk R Kanter, MD, Principal Investigator — Children's Healthcare of Atlanta, Pediatric Surgery
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States